CLINICAL TRIAL: NCT07172724
Title: "First-in-human, Phase 1, Double-blind, Randomized, Placebo-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of the Vivaxin Vaccine for Malaria Caused by Plasmodium Vivax."
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of the Vivaxin Vaccine for Malaria Caused by Plasmodium Vivax."
Acronym: Vivaxin-001
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: University of Sao Paulo (Other); Financiadora de Estudos e Projetos (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); INCTV National Institute of Vaccine Science and Technology (Unknown); The Ministry of Science, Technology and Innovation, Brazil (Unknown); CT Vacinas - Centro de Tecnologia em Vacinas/Universidade Federal de Minas Gerais (Unknown)
Responsible Party: Principal Investigator, Helton da Costa Santiago, Study Director, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Vivaxin-001; U1111-1321-7560 (Other: WHO International Clinical Trials Registry Plataforms); 89852825.0.0000.0444 (Other: Plataforma Brasil); 7.783.109 (Other: Ethics Committee of the Federal University of Minas Gerais/Campus Saude)
Record Dates: First submitted 2025-08-19; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Malaria Vivax
Keywords: vaccine; malaria; Plasmodium vivax; prevention; malaria vivax
MeSH Terms: conditions — Malaria, Vivax; Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 - 25 µg of Vivaxin (Experimental): Twelve healthy participants of both sexes, aged 18 to 59 years, with no prior exposure to malaria will receive three doses of 25 µg of Vivaxin, with 28-day intervals between doses.
  Interventions: Biological: Vivaxin vaccine manufactured by CT Vacinas/Cristália Laboratory
- Arm 2 - 50 µg of Vivaxin (Experimental): Twelve healthy participants of both sexes, aged 18 to 59 years, with no prior exposure to malaria will receive three doses of 50 µg of Vivaxin, with 28-day intervals between doses.
  Interventions: Biological: Vivaxin vaccine manufactured by CT Vacinas/Cristália Laboratory
- Arm 3 - 100 µg of Vivaxin (Experimental): Twelve healthy participants of both sexes, aged 18 to 59 years, with no prior exposure to malaria will receive three doses of 100 µg of Vivaxin, with 28-day intervals between doses.
  Interventions: Biological: Vivaxin vaccine manufactured by CT Vacinas/Cristália Laboratory
- Placebo (Placebo Comparator): Four healthy participants of both sexes, aged 18 to 59 years, with no prior exposure to malaria will receive three doses of placebo, with 28-day intervals between doses.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Vivaxin vaccine manufactured by CT Vacinas/Cristália Laboratory — lyophilized antigen for reconstitution with the adjuvant CTVad (a squalene-based nanoemulsion), at the time of use.
  Arms: Arm 1 - 25 µg of Vivaxin; Arm 2 - 50 µg of Vivaxin; Arm 3 - 100 µg of Vivaxin
Other: Placebo — adjuvant CTVad (a squalene-based nanoemulsion)
  Arms: Placebo

SUMMARY:
Phase 1 clinical trial to evaluate the safety, reactogenicity, and immunogenicity of a malaria vaccine named Vivaxin against the protozoan Plamodium vivax in participants with no prior malaria infection

DETAILED DESCRIPTION:
Vivaxin is being developed for use as a prophylactic vaccine against malaria caused by Plasmodium vivax, the dominant species in Brazil.

The study will consist of the assessment of the safety, reactogenicity, and immunogenicity of the vaccine following intramuscular administration of three doses of 0.3 mL/dose, with a 28-day interval between each dose, in healthy participants of both sexes, aged 18 to 59 years, with no prior exposure to malaria.

This will be a Phase 1, first-in-human, randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety and immunogenicity of the investigational product, Vivaxin vaccine.

A total of 16 participants will be included in each of the 3 study arms, based on Vivaxin dose levels: 25 µg, 50 µg, and 100 µg. In each arm, 12 participants will receive the Vivaxin vaccine, and 4 participants will receive a placebo. Additionally, a sentinel cohort will be included within each arm:

Arm 1 - 25 µg of Vivaxin (N=12) or placebo (N=4):

Twelve participants will receive three doses of 25 µg of Vivaxin, with 28-day intervals between doses, and four participants will receive three doses of placebo, also at 28-day intervals. The first four individuals enrolled will comprise the sentinel group. Three of these will receive Vivaxin and one will receive placebo, randomized in a blinded manner. They will be observed for at least 7 days prior to proceeding with vaccination of the remaining participants in this arm. Vaccination of the remaining participants will proceed only after confirming that no study-halting criteria have been met.

Arm 2 - 50 µg of Vivaxin (N=12) or placebo (N=4):

Twelve participants will receive three doses of 50 µg of Vivaxin, with 28-day intervals, and four participants will receive placebo under the same schedule. The first four individuals enrolled will comprise the sentinel group (three receiving Vivaxin, one receiving placebo). They will be observed for at least 7 days before vaccination continues in this arm. Continuation is contingent upon confirmation that no halting criteria have been met.

Arm 3 - 100 µg of Vivaxin (N=12) or placebo (N=4):

Twelve participants will receive three doses of 100 µg of Vivaxin, spaced 28 days apart, and four participants will receive placebo at the same intervals. As with the other arms, the first four individuals enrolled will form the sentinel group and will be observed for at least 7 days before vaccination of the remaining participants in the arm is permitted, conditional on the absence of any study-halting criteria.

All participants in the sentinel cohorts will be observed at the research center for 60 minutes post-vaccination (vaccine or placebo). All other participants will be observed for a minimum of 30 minutes. All participants will be followed for 360 days with regular clinical assessments, including:

Telephone follow-ups on Days 1 and 3 (post-first dose), Days 29 and 31 (1 and 3 days post-second dose), Days 57 and 59 (1 and 3 days post-third dose), and monthly thereafter until study completion;

In-person visits on Days 7 and 14 (1 and 2 weeks post-first dose), Day 28 (second dose), Days 35 and 42 (1 and 2 weeks post-second dose), Day 56 (third dose), Days 63 and 70 (1 and 2 weeks post-third dose), and Days 84, 120, 180, 270, and 360 post-vaccination (end of study).

Participants will be sequentially enrolled and allocated to Arms 1, 2, and 3 of the study, receiving 25 µg, 50 µg, and 100 µg of the investigational product, respectively. In each arm, 12 participants will receive the Vivaxin vaccine and 4 participants will receive placebo, totaling 16 participants per arm.

The first four randomized individuals in each arm will comprise the sentinel group and will be observed for at least 7 days prior to continuation of vaccination in that arm. Adverse events (AEs) from each sentinel cohort will be reviewed by the Protocol and Safety Review Team (PSRT) within 7 days following vaccination. If no halting criteria are met, vaccination of the remaining participants in the arm will proceed.

After the first 14 days of follow-up of all participants in Arm 1, a blinded safety review will be conducted by the PSRT to determine whether dose escalation may proceed. If no halting criteria are observed, the PSRT will recommend study continuation. Should any halting criteria be met or any PSRT member deem it necessary, a meeting with the Independent Data and Safety Monitoring Committee (DSMC) will be convened. The DSMC, upon review of the safety data, may recommend continuation as planned, propose protocol modifications, or advise study suspension. This procedure will be repeated at each dose escalation stage.

If the PSRT recommends proceeding, participants in Arm 2 (50 µg) will be vaccinated, beginning with the sentinel cohort of four individuals who will be observed for 7 days before continued randomization in the arm. Meanwhile, Arm 1 may continue with second and third immunizations, observing the sentinel group of each dose for 7 days prior to proceeding with full-arm administration.

Upon completion of the first 14 days of follow-up in Arm 2, a safety analysis will be conducted by the PSRT to determine whether escalation to Arm 3 may proceed. As with the previous arms, the first four individuals in Arm 3 will form the sentinel group and will be observed for 7 days prior to continued vaccination in that arm.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant women and men aged between 18 and 59 years;
2. Willingness to participate in the study and undergo all study procedures, as demonstrated by signing the informed consent form (ICF);
3. In good general health, as determined by medical examination;
4. Women of childbearing potential must agree to use an acceptable* contraceptive method for at least 30 days prior to the first vaccination and for at least 6 months following administration of the first dose of the investigational product, ensuring at least 3 months after the final vaccine dose have elapsed;
5. Agreement not to donate blood during the course of study participation.

   * Acceptable contraceptive methods:

     * Barrier methods, including condom or cervical cap;
     * Surgically sterile partner/participant (including those who have undergone vasectomy, hysterectomy, bilateral oophorectomy, and/or tubal ligation) who is the sole sexual partner;
     * Intrauterine device (with or without hormones);
     * Hormonal birth control methods (oral, topical, injectable, or implantable);
     * True sexual abstinence that is consistent with the participant's preferred and usual lifestyle.

Note: Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) or withdrawal (coitus interruptus) will not be considered acceptable methods.

Exclusion Criteria:

1. Prior history of malaria infection confirmed by serological testing;
2. Prior history of malaria vaccination;
3. Intention to travel to a malaria-endemic area during the study period;
4. Pregnant or breastfeeding women, or those intending to become pregnant or breastfeed within the first 6 months of the study;
5. Evidence of clinically active disease, such as but not limited to: neurological, renal, cardiovascular, endocrine, pulmonary, hepatic, hematological, immunological, neoplastic, or infectious diseases;
6. Use of concomitant medication for control of an underlying medical condition;
7. Positive serological test for HBV, HCV, or HIV;
8. Any condition that, in the opinion of the study investigator, could pose a risk to the participant or confound the study results, including clinically stable chronic conditions such as diabetes, hypertension, or neuralgias, among others;
9. Psychiatric illness or cognitive impairment that, in the opinion of the investigator, may affect the participant's ability to comply with the clinical study schedule;
10. History of alcohol or substance abuse within 12 months prior to enrollment that resulted in family, medical, or occupational problems;
11. History of severe allergic reaction or anaphylaxis to any component of the vaccine;
12. History of asplenia;
13. Participation in any other investigational clinical trial within 12 months prior to inclusion in this study;
14. Plans to participate in other clinical trials concurrently with this study;
15. Use of any immunosuppressive therapy within 3 months prior to enrollment or plans to use such therapy within 3 months after vaccination, including corticosteroids or other immunosuppressive drugs. An immunosuppressive dose of corticosteroid is defined as the equivalent of 20 mg/day of prednisone for more than one week. Topical or nasal corticosteroids are not considered immunosuppressive;
16. Use of blood products (including blood or immunoglobulins) within 3 months prior to enrollment in this study, or plans to use them during the study period;
17. Suspected or confirmed fever (axillary temperature ≥ 37.8 °C) within 72 hours prior to study enrollment. Enrollment should be postponed until the participant has been afebrile for at least 72 hours;
18. Receipt of any live attenuated or inactivated vaccine within 28 or 14 days, respectively, prior to administration of the investigational product, or plans for immunization within 28 days after enrollment in the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety and reactogenicity of adverse events (AE) in the first 14 days | Day 14 after each immunization
  Frequency and intensity of solicited AEs with a possible causal relationship or higher up to 14 days after intramuscular administration of Vivaxin vaccine.
Safety and reactogenicity of EA in the first 28 days | Day 28 after each immunization
  Frequency and intensity of unsolicited AEs with a possible causal relationship or higher up to 28 days after intramuscular administration of Vivaxin vaccine.
Safety and reactogenicity of serious AEs (SAEs) and AEs of special interest (AESI) throughout the study duration | through study completion, an average of 18 months
  Frequency and intensity of SAEs and AESIs throughout the study duration after intramuscular administration of Vivaxin vaccine.
Dose selection | Day 28 after the third dose of the vaccine of all participants
  Selection of a safe and immunogenic dose of Vivaxin to continue clinical development.

SECONDARY OUTCOMES:
Levels of IgG antibodies | Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 120, 180, 270 and 360 after immunization
  Mean levels of IgG antibodies, calculated by the geometric mean of the titers against vaccine and parasitic antigens on days 7, 14, 28, 35, 42, 56, 63, 70, 84, 120, 180, 270 and 360 in relation to time 0 and placebo, by ELISA.

OTHER OUTCOMES:
Levels of IgM, IgG1, IgG2, IgG3, IgG4 and IgA against vaccine and parasitic antigens | Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 120, 180, 270 and 360 after immunization
  1.Levels of IgM, IgG1, IgG2, IgG3, IgG4 and IgA against vaccine and parasitic antigens, such as the three variants of the Plasmodium vivax circumsporozoite protein (PvCSP), after intramuscular administration of the Vivaxin vaccine, in relation to time 0 and placebo, by ELISA.
Observe the multifunctional cellular immune response by evaluating the quality and frequency of CD4+ and CD8+ T lymphocytes in response to vaccine and parasite antigens | Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 120, 180, 270 and 360 after immunization
  Frequency and quality of CD4+ and CD8+ T lymphocytes that produce multiple cytokines (such as IFNγ, IL-4/IL-13, IL-17, TNFa and IL-10) in response to vaccine and parasite antigens, on days 7, 14, 28, 35, 42, 56, 63, 70, 84, 120, 180, 270 and 360 after intramuscular administration of the Vivaxin vaccine, in relation to time 0 and placebo, by ELISA
Levels of IFNγ and other cytokines | Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 120, 180, 270 and 360 after immunization
  Levels of IFNγ and other cytokines (in pg/mL) produced by peripheral blood mononuclear cells (PBMC) in culture in response to vaccine and parasite antigens on days 7, 14, 28, 35, 42, 56, 63, 70, 84, 120, 180, 270 and 360 after intramuscular administration of Vivaxin vaccine, in relation to time 0 and placebo, by ELISA.
Observe the genomic and transcriptomic diversity to better understand the immune response to the vaccine | through study completion, an average of 18 months
  Contribution of genomic and transcriptomic diversity to safety, reactogenicity and adverse event profile, as well as to the characterization of the humoral and cellular immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo T Gazzinelli, DVM, PhD, Study Chair — Vaccine Technology Center (CT Vacinas)
Locations (1):
- Centro de Pesquisas Clínicas (CPC) do Hospital das Clínicas (HC) da UFMG/ Filial Ebserh, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We are currently assessing the feasibility of sharing IPD, considering ethical, legal, and institutional requirements. A final decision has not yet been made.

REFERENCES:
- See also: World Malaria Report 2024 — https://www.who.int/teams/global-malaria-programme/reports/world-malaria-report-2024
- See also: Malaria Day in the Americas - an overview of malaria in Brazil in 2022 and the first half of 2023 — https://www.gov.br/saude/pt-br/centrais-de-conteudo/publicacoes/boletins/epidemiologicos/edicoes/2024/boletim-epidemiologico-volume-55-no-01/view